CLINICAL TRIAL: NCT05789251
Title: Assess the Possibility of Diagnosing Diabetes and Rediabetes Following Oral Induced Hyperglycemia in Patients With Dunnigan's Partial Familial Lipodystrophy by Replacing 75 g of Glucose With a Standardized Carbohydrate Breakfast and Continuous Interstitial Monitoring Glucose)
Acronym: HGPO-DUN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/CHU/03
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Lipodystrophy
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standardized breakfast to replace in fine oral induced hyperglycemia test (Experimental): Standardized breakfast to replace in fine oral induced hyperglycemia test
  Interventions: Diagnostic Test: Standardized breakfast

INTERVENTIONS:
Diagnostic Test: Standardized breakfast — Standardized breakfast to replace in fine oral induced hyperglycemia test

SUMMARY:
Dunnigan's syndrome is a partial familial lipodystrophy due to a mutation in the Lamine A LMNA gene. This very rare syndrome is 20 times more common in Réunion compared to the rest of Europe with several families suffering from a unique variant of LMNA, the p.(Thr655Asnfs*49) variant known as the "Reunion variant", the appearance of which in Reunion dates back to the 17th century. This variant is expressed in homozygous and heterozygous form and has only been identified in subjects from Reunion. Clinically, patients with Dunnigan's have an absence of subcutaneous fatty tissue which mainly affects the lower part of the body and leads to severe insulin resistance responsible for early diabetes. To detect these metabolic complications as early as possible, an annual follow-up of the subjects is recommended with the performance of an OGTT test annually in non-diabetic subjects. This problem is identical for patients with cystic fibrosis leading to the same recommendation. However, whether in our experience of monitoring patients with Dunningan's lipodystrophy, in subjects at risk of diabetes or in subjects with cystic fibrosis, the OGTT test and even more so its repetition is poorly accepted, which can lead to lack of patient follow-up. An alternative solution to the OGTT is therefore justified.

In the literature, different avenues have been explored. First, given oral glucose intolerance, replacement with a standardized breakfast has been explored in several studies. Another alternative tested in the population of subjects with cystic fibrosis is the use of an interstitial glucose sensor for screening for carbohydrate abnormalities.

In view of the literature, we formulate several hypotheses that will be tested in our study:

1. The intake of a standardized breakfast containing 75g of carbohydrates is comparable to the ingestion of 75g of glucose on the result of the OGTT test at 120 min for the diagnosis of carbohydrate abnormalities (diabetes and prediabetes) in patients with Dunnigan's lipodystrophy.
2. The continuous recording of interstitial glycaemia over several days allows the diagnosis of glucidic abnormalities equivalent to the classic OGTT in this population; possibly by identifying glycemic variations not seen by a single OGTT test. Thus the installation of an interstitial sensor over several days could be an alternative to the realization of the OGTT in the identification of carbohydrate disorders in patients with Dunnigan's lipodystrophy.
3. There will be a similar profile but a time lag between venous glycemic curves and interstitial blood glucose measurements after OGTT.
4. Replacing the oral glucose load of the classic OGTT (gold standard) with a standardized carbohydrate breakfast leads to similar interstitial glycaemia curves but with a time lag.

ELIGIBILITY:
Inclusion Criteria:

* Subject with Dunnigan's partial familial lipodystrophy followed at Reunion University Hospital not known to be diabetic.

Aged 18 to 75 Having given their informed consent.

Exclusion Criteria:

* Diabetic patient Patient scheduled for scan within 7 days of freestyle placement protected persons: "pregnant woman, parturient, nursing mother, person deprived of liberty by judicial or administrative decision, minor, and person subject to a measure of legal protection: guardianship or curatorship)"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
standardized breakfast test resuslt compare to oral induced hyperglycemia test | 2 hours after standardized breakfast
  To assess the concordance between the standard breakfast-induced hyperglycemia test and the classic oral induced hyperglycemia test (gold standard) on the diagnosis of glycemic abnormalities at 120 minutes (min) in patients with Dunnigan's Lipodystrophy in Reunion. It is considered good if > 80%

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de La Réunion, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: No